CLINICAL TRIAL: NCT02173054
Title: An Evaluator-blind, Randomized, Vehicle-controlled Efficiency of Adjunctive Usage of a Moisturizer Containing Licochalcone A, L-carnitine and 1,2-decanediol With Adapalene Gel for Improvement of Local Tolerance in Thai Acne Subjects
Brief Title: An Efficiency of a Moisturizer Containing Licochalcone A, L-carnitine and 1,2-decanediol With Adapalene Gel in Acne
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Acne and adjuctive moisturizer
Record Dates: First submitted 2014-06-18; First posted 2014-06-24 (Estimated); Results first posted 2016-02-26 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2016-11

CONDITIONS: Acne
Keywords: Acne; Moisturizer; Efficacy; Irritation
MeSH Terms: conditions — Acne Vulgaris | interventions — eucerin; licochalcone A; Carnitine; Adapalene

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Adapalene gel (Placebo Comparator): Evening
  * Wash face by prepared facial foam and dry your face
  * Apply adapalene gel all over the face
  Interventions: Other: Adapalene gel
- Adapalene gel with placebo moisturizer (Placebo Comparator): Morning
  * Wash face by prepared facial foam and dry their face
  * Apply placebo cream all over the face
  Evening
  * Wash face by prepared facial foam and dry your face
  * Apply adapalene gel all over the face
  * Apply placebo cream all over the face
  Interventions: Other: Adapalene gel with placebo moisturizer
- Adapalene gel with Eucerin (Active Comparator): Morning
  * Wash face by prepared facial foam and dry their face
  * Apply Eucerin cream all over the face
  Evening
  * Wash face by prepared facial foam and dry your face
  * Apply adapalene gel all over the face
  * Apply Eucerin cream all over the face
  Interventions: Other: Adapalene gel with Eucerin

INTERVENTIONS:
Other: Adapalene gel with Eucerin — Eucerin: 2 fingertip unit to cover all over the face twice a day. Adapalene gel: 2 fingertip unit to cover all over the face before going to bed
  Other Names: licochalcone A + L-carnitine + decanediol (Eucerin); Adapalene gel (Differin)
  Arms: Adapalene gel with Eucerin
Other: Adapalene gel — Adapalene gel: 2 fingertip unit to cover all over the face before going to bed
  Other Names: Adapalene gel (Differin)
  Arms: Adapalene gel
Other: Adapalene gel with placebo moisturizer — Placebo: 2 fingertip unit to cover all over the face twice a day. Adapalene gel: 2 fingertip unit to cover all over the face before going to bed
  Other Names: •Adapalene gel (Differin)
  Arms: Adapalene gel with placebo moisturizer

SUMMARY:
Acne is an inflammation of sebaceous glands and follicles. Applying topical treatments such as adapalene gel may cause irritant adverse effects. Hence, using a moisturizer is another way to protect or relieve this undesirable event. Moisturizers that have anti-inflammatory property could reduce irritant effects, emergent from using topical treatment and also reduce severity of acne.

Research teams chose an adapalene gel to act as topical treatment for curing acne. It has anti-inflammatory and comedolytic effects and has fewer side effects than other groups of topical retinoic acids. However, peeling skin, redness skin, tingling sensation or itching sensation may occur if they are continually used for a long period. Thus, for the purpose of studying the efficacy of moisturizer containing licochalcone A, L-carnitine and 1,2-decanediol in reducing irritant effect of using adapalene gel (Licochalcone A has anti-inflammatory effect, L-carnitine decrease sebum production and 1,2-decanediol has anti-bacterial effect).

DETAILED DESCRIPTION:
The investigators team research with patients by separate patients into 3 groups and compare among each other. In the first group use only adapalene gel, the second group use adapalene gel with moisturizer containing three substances mentioned above, and the last group use adapalene gel with placebo moisturizer. To compare outcomes among 3 groups, the investigators will measure degree of redness, scale, oily face, moist, number of acne, quality of life, and satisfaction after using moisturizer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years old or above
2. Participants have to control the birth for example, condom method, intrauterine device method before participate in the research at least 1 month until 6 months after research finish.
3. being diagnosed acne vulgaris by dermatologist in mild to moderate degree based on Investigators' Global Assessment scale of FDA

Exclusion Criteria:

1. Use oral or injected antibiotics or other oral medicine treating acne for example, isotretinoin, oral contraceptives, or spironolactone group during 4 weeks before participate this research
2. Have other active skin diseases at face during 2 weeks before participate the research
3. Allergic to adapalene gel and moisturizer
4. Have severe or uncontrolled underlying diseases
5. Getting pregnant or during breast feeding
6. Other types of acne(not acne vulgaris)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-07; Primary Completion 2015-02 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Papapit Tuchinda, MD, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital Mahidol Univeristy, Bangkok, Bangkok, Thailand

REFERENCES:
- [Derived] Chularojanamontri L, Tuchinda P, Kulthanan K, Varothai S, Winayanuwattikun W. A double-blinded, randomized, vehicle-controlled study to access skin tolerability and efficacy of an anti-inflammatory moisturizer in treatment of acne with 0.1% adapalene gel. J Dermatolog Treat. 2016;27(2):140-5. doi: 10.3109/09546634.2015.1079298. Epub 2015 Sep 2. PMID 26293170

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period: between June 2014 and December 2014 Location: Department of Dermatology, Siriraj Hospital, Mahidol University, Thailand
Groups:
- Adapalene Gel: Evening
  * Wash face by prepared facial foam and dry your face
  * Apply adapalene gel all over the face
  Adapalene gel: Adapalene gel: 2 fingertip unit to cover all over the face before going to bed
- Adapalene Gel With Placebo Moisturizer: Morning
  * Wash face by prepared facial foam and dry their face
  * Apply placebo cream all over the face
  Evening
  * Wash face by prepared facial foam and dry your face
  * Apply adapalene gel all over the face
  * Apply placebo cream all over the face
  Adapalene gel with placebo moisturizer: Placebo: 2 fingertip unit to cover all over the face twice a day.
  Adapalene gel: 2 fingertip unit to cover all over the face before going to bed
- Adapalene Gel With Eucerin: Morning
  * Wash face by prepared facial foam and dry their face
  * Apply Eucerin cream all over the face
  Evening
  * Wash face by prepared facial foam and dry your face
  * Apply adapalene gel all over the face
  * Apply Eucerin cream all over the face
  Adapalene gel with Eucerin: Eucerin: 2 fingertip unit to cover all over the face twice a day.
  Adapalene gel: 2 fingertip unit to cover all over the face before going to bed
Period: Overall Study
Arm/Group | Adapalene Gel | Adapalene Gel With Placebo Moisturizer | Adapalene Gel With Eucerin
Started | 40 | 40 | 40
Completed | 39 | 40 | 39
Not Completed | 1 | 0 | 1
Not completed — lack of compliance | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adapalene Gel | Adapalene Gel With Placebo Moisturizer | Adapalene Gel With Eucerin | Total
Number analyzed (Participants) | 40 | 40 | 40 | 120
Age, Continuous [Mean (Full Range); unit: years] | 27.3 [19 to 43] | 27.2 [20 to 40] | 28.1 [18 to 49] | 27.5 [18 to 49]
Gender [Count of Participants; unit: Participants]
  Female | 22 | 19 | 26 | 67
  Male | 18 | 21 | 14 | 53
Region of Enrollment [Number; unit: participants]
  Thailand | 40 | 40 | 40 | 120

OUTCOME MEASURES:

1. Primary Outcome: Reduction of Undesirable Effects
Description: * Undesirable effects were evaluated from skin's condition/signs(erythema, dryness and scaling) are evaluated by dermatologist. (none; mild; moderate; severe) and subject interview/symptoms(stinging/burning and pruritis) are evaluated by participants.(none; mild; moderate; severe). There were assessed at 2nd week, 4th week, and 8th week.
  * The worst score of each parameter which was defined as the worst local tolerance score is demonstrated and compared among 3 groups as shown.
Time Frame: 2nd week, 4th week, and 8th week
Population: The reasons for drop out were lack of compliance (n=1, group A: adapalene gel alone) and consent withdrawal at patient's request (n=1, group C: adapalene with Eucerin)
Measure: Number; unit: participants
Arm/Group | Adapalene Gel | Adapalene Gel With Placebo Moisturizer | Adapalene Gel With Eucerin
Number analyzed (Participants) | 39 | 40 | 39
participants
  Erythema (none) | 26 | 38 | 35
  Erythema (mild) | 10 | 2 | 4
  Erythema (moderate) | 3 | 0 | 0
  Dryness (none) | 21 | 29 | 32
  Dryness (mild) | 14 | 11 | 6
  Dryness (moderate) | 4 | 0 | 1
  Scaling (none) | 13 | 16 | 24
  Scaling (mild) | 22 | 24 | 14
  Scaling (moderate) | 4 | 0 | 1
  Stinging (none) | 6 | 9 | 6
  Stinging (mild) | 14 | 12 | 11
  Stinging (moderate) | 10 | 13 | 13
  Stinging (severe) | 9 | 6 | 9
  Pruritus (none) | 18 | 21 | 23
  Pruritus (mild) | 10 | 8 | 9
  Pruritus (moderate) | 7 | 6 | 5
  Pruritus (severe) | 4 | 5 | 2
Statistical Analysis 1: Comparison: Adapalene Gel vs Adapalene Gel With Placebo Moisturizer vs Adapalene Gel With Eucerin; Test type: Superiority or Other; p = 0.001, Kruskal-Wallis — This statistical analysis was used to compare number of participants who had erythema among 3 groups
Statistical Analysis 2: Comparison: Adapalene Gel vs Adapalene Gel With Placebo Moisturizer vs Adapalene Gel With Eucerin; Test type: Superiority or Other; p = 0.016, Kruskal-Wallis — This statistical analysis was used to compare number of participants who had dryness among 3 groups
Statistical Analysis 3: Comparison: Adapalene Gel vs Adapalene Gel With Placebo Moisturizer vs Adapalene Gel With Eucerin; Test type: Superiority or Other; p = 0.025, Kruskal-Wallis — This statistical analysis was used to compare number of participants who had scaling among 3 groups
Statistical Analysis 4: Comparison: Adapalene Gel vs Adapalene Gel With Placebo Moisturizer vs Adapalene Gel With Eucerin; Test type: Superiority or Other; p = 0.571, Kruskal-Wallis — This statistical analysis was used to compare number of participants who had stinging among 3 groups
Statistical Analysis 5: Comparison: Adapalene Gel vs Adapalene Gel With Placebo Moisturizer vs Adapalene Gel With Eucerin; Test type: Superiority or Other; p = 0.449, Kruskal-Wallis — This statistical analysis was used to compare number of participants who had pruritus among 3 groups

2. Secondary Outcome: Reduction of Severity of Acne
Description: * Evaluation from mean counts of inflammatory, noninflammatory, and total acne lesions at baseline, and at 2, 4, and 8 weeks
  * Total acne lesions = inflammatory + noninflammatory acne lesions
  * Reduction of lesions counts are considered to be a better outcome
Time Frame: baseline, 2nd week, 4th week and 8th week
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Adapalene Gel | Adapalene Gel With Placebo Moisturizer | Adapalene Gel With Eucerin
Number analyzed (Participants) | 39 | 40 | 39
Lesions
  Baseline Total Lesion Count | 35.9 (49.1) | 27.4 (37.0) | 25.5 (16.9)
  Week 2 Total Lesion Count | 41 (65.7) | 26.6 (29.3) | 23.8 (16.6)
  Week 4 Total Lesion Count | 39 (54.2) | 27.3 (25.2) | 25.7 (16.7)
  Week 8 Total Lesion Count | 28.9 (33.3) | 26.8 (22.5) | 19.9 (15.2)
  Baseline Inflammatory Lesion Counts | 3.5 (3.9) | 3 (2.6) | 3.8 (3.3)
  Week 2 Inflammatory Lesion Counts | 4.5 (6.6) | 4.1 (7.4) | 3.6 (3.9)
  Week 4 Inflammatory Lesion Counts | 3.6 (5.4) | 2.9 (2.9) | 3.4 (3.5)
  Week 8 Inflammatory Lesion Counts | 2.5 (5.6) | 3.1 (4.1) | 2.4 (3.0)
  Baseline Noninflammatory Counts | 32.4 (48.0) | 24.5 (37.3) | 21.6 (16.2)
  Week 2 Noninflammatory Counts | 36.5 (61.9) | 22.5 (28.1) | 20.5 (15.3)
  Week 4 Noninflammatory Counts | 35.4 (50.6) | 24.4 (24.4) | 22.6 (16.1)
  Week 8 Noninflammatory Counts | 26.4 (29.1) | 23.7 (20.1) | 17.7 (14.7)
Statistical Analysis 1: Comparison: Adapalene Gel; Test type: Superiority or Other; p = 0.059, wilcoxan signed ranks test — This statistical analysis was used to evaluate the change in total lesion counts at baseline and 8th week
Statistical Analysis 2: Comparison: Adapalene Gel With Placebo Moisturizer; Test type: Superiority or Other; p = 0.697, wilcoxan signed ranks test — This statistical analysis was used to evaluate the change in total lesion counts at baseline and 8th week
Statistical Analysis 3: Comparison: Adapalene Gel With Eucerin; Test type: Superiority or Other; p = 0.028, wilcoxan signed ranks test — This statistical analysis was used to evaluate the change in total lesion counts at baseline and 8th week
Statistical Analysis 4: Comparison: Adapalene Gel; Test type: Superiority or Other; p = 0.001, wilcoxan signed ranks test — This statistical analysis was used to evaluate the change in inflammatory lesion counts at baseline and 8th week
Statistical Analysis 5: Comparison: Adapalene Gel With Placebo Moisturizer; Test type: Superiority or Other; p = 0.755, wilcoxan signed ranks test — This statistical analysis was used to evaluate the change in inflammatory lesion counts at baseline and 8th week
Statistical Analysis 6: Comparison: Adapalene Gel With Eucerin; Test type: Superiority or Other; p = 0.003, wilcoxan signed ranks test — This statistical analysis was used to evaluate the change in inflammatory lesion counts at baseline and 8th week
Statistical Analysis 7: Comparison: Adapalene Gel; Test type: Superiority or Other; p = 0.205, wilcoxan signed ranks test — This statistical analysis was used to evaluate the change in non inflammatory lesion counts at baseline and 8th week
Statistical Analysis 8: Comparison: Adapalene Gel With Placebo Moisturizer; Test type: Superiority or Other; p = 0.576, wilcoxan signed ranks test — This statistical analysis was used to evaluate the change in non inflammatory lesion counts at baseline and 8th week
Statistical Analysis 9: Comparison: Adapalene Gel With Eucerin; Test type: Superiority or Other; p = 0.160, wilcoxan signed ranks test — This statistical analysis was used to evaluate the change in non inflammatory lesion counts at baseline and 8th week

3. Primary Outcome: Skin Tolerability: Skin Sebum Content and Skin Hydration
Description: Skin tolerability was assessed by measuring the skin surface sebum content, skin hydration with the Sebumeter SM815 and Corneometer CM825, respectively
Time Frame: Skin tolerability was assessed at baseline and week 8. The changes of skin tolerability between baseline and 8th week of the 3 groups were compared.
Measure: Mean (Standard Deviation); unit: µg/cm^2
Arm/Group | Adapalene Gel | Adapalene Gel With Placebo Moisturizer | Adapalene Gel With Eucerin
Number analyzed (Participants) | 39 | 40 | 39
µg/cm^2
  Baseline Sebumeter | 75.7 (34.4) | 71.2 (42.4) | 73.7 (31.2)
  Week 8 Sebumeter | 63.6 (31.7) | 59.9 (55.3) | 64.2 (35.0)
  Baseline Corneometer | 51.7 (10.0) | 50.2 (10.5) | 46.7 (11.3)
  Week 8 Corneometer | 50.9 (10.9) | 49.5 (9.4) | 48.6 (9.3)
Statistical Analysis 1: Comparison: Adapalene Gel; Test type: Superiority or Other; p = 0.078, Paired t-test — This statistical analysis was used to evaluate the change in skin sebum content at baseline and 8th week of the Adapalene gel group
Statistical Analysis 2: Comparison: Adapalene Gel With Placebo Moisturizer; Test type: Superiority or Other; p = 0.167, Paired t-test — This statistical analysis was used to evaluate the change in skin sebum content at baseline and 8th week of the Adapalene gel with placebo moisturizer group
Statistical Analysis 3: Comparison: Adapalene Gel With Eucerin; Test type: Superiority or Other; p = 0.134, Paired t-test — This statistical analysis was used to evaluate the change in skin sebum content at baseline and 8th week of the Adapalene gel with Eucerin group
Statistical Analysis 4: Comparison: Adapalene Gel; Test type: Superiority or Other; p = 0.978, Paired t-test — This statistical analysis was used to evaluate the change in skin hydration at baseline and 8th week of the Adapalene gel group
Statistical Analysis 5: Comparison: Adapalene Gel With Placebo Moisturizer; Test type: Superiority or Other; p = 0.273, Paired t-test — This statistical analysis was used to evaluate the change in skin hydration at baseline and 8th week of the Adapalene gel with placebo moisturizer group
Statistical Analysis 6: Comparison: Adapalene Gel With Eucerin; Test type: Superiority or Other; p = 0.735, Paired t-test — This statistical analysis was used to evaluate the change in skin hydration at baseline and 8th week of the Adapalene gel with Eucerin group

4. Primary Outcome: Skin Tolerability: Transepidermal Water Loss (TEWL)
Description: Skin tolerability was assessed by measuring TEWL with the Tewameter TM300
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: g/m^2h
Arm/Group | Adapalene Gel | Adapalene Gel With Placebo Moisturizer | Adapalene Gel With Eucerin
Number analyzed (Participants) | 39 | 40 | 39
g/m^2h
  Baseline TEWL | 9.8 (3.3) | 10.4 (4.6) | 10.6 (3.7)
  Week 8 TEWL | 12.3 (4.8) | 11.8 (5.4) | 11.5 (3.3)
Statistical Analysis 1: Comparison: Adapalene Gel; Test type: Superiority or Other; p = 0.0002, Paired t-test — This statistical analysis was used to evaluate the change in TEWL at baseline and 8th week of the Adapalene gel group
Statistical Analysis 2: Comparison: Adapalene Gel With Placebo Moisturizer; Test type: Superiority or Other; p = 0.007, Paired t-test — This statistical analysis was used to evaluate the change in TEWL at baseline and 8th week of the Adapalene gel with placebo moisturizer group
Statistical Analysis 3: Comparison: Adapalene Gel With Eucerin; Test type: Superiority or Other; p = 0.123, Paired t-test — This statistical analysis was used to evaluate the change in TEWL at baseline and 8th week of the Adapalene gel with Eucerin group

5. Secondary Outcome: Reduction of Severity of Acne: Acne Severity Index (ASI)
Description: * The ASI score was calculated from the number of papules + (2 x pustules) + (comedones/4)
  * Decrease of ASI score are considered to be a better outcome
Time Frame: baseline, 2nd week, 4th week and 8th week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adapalene Gel | Adapalene Gel With Placebo Moisturizer | Adapalene Gel With Eucerin
Number analyzed (Participants) | 39 | 40 | 39
units on a scale
  Baseline ASI | 11.7 (13.6) | 9.4 (9.5) | 9.5 (5.8)
  Week 2 ASI | 14.4 (20.8) | 10.4 (11.3) | 8.7 (6.1)
  Week 4 ASI | 13.6 (19.4) | 9.2 (7.5) | 9.2 (5.9)
  Week 8 ASI | 9.5 (13.7) | 9.3 (8.5) | 7.1 (5.3)
Statistical Analysis 1: Comparison: Adapalene Gel; Test type: Superiority or Other; p = 0.005, wilcoxan signed ranks test — This statistical analysis was used to evaluate the change in ASI score at baseline and 8th week
Statistical Analysis 2: Comparison: Adapalene Gel With Placebo Moisturizer; Test type: Superiority or Other; p = 0.606, wilcoxan signed ranks test — This statistical analysis was used to evaluate the change in ASI score at baseline and 8th week
Statistical Analysis 3: Comparison: Adapalene Gel With Eucerin; Test type: Superiority or Other; p = 0.001, wilcoxan signed ranks test — This statistical analysis was used to evaluate the change in ASI score at baseline and 8th week

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Adapalene Gel | Adapalene Gel With Placebo Moisturizer | Adapalene Gel With Eucerin
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No